CLINICAL TRIAL: NCT03050398
Title: A Companion Sample Collection Protocol to Support the Discovery of Breast Cancer Aberrations With Treatment of CDK4/6 Therapy/LEE011/Ribociclib
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: GCP issues.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLEE011AUS42
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: HR-positive; HER2-negative; Advanced breast cancer; LEE011; ribociclib; letrozole; femara; CDK; CDK4; CDK6; CDK4/6; CDK4/6 inhibitor; Phase III; Phase IIIb; ER-positive; PR-positive; Postmenopausal; Premenopausal; Men
MeSH Terms: conditions — Breast Neoplasms; Multiple Endocrine Neoplasia Type 1 | interventions — ribociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ribociclib + letrozole (Experimental): ribociclib with letrozole per the core study
  Interventions: Drug: Ribociclib; Drug: letrozole

INTERVENTIONS:
Drug: Ribociclib — ribociclib + letrozole
Drug: letrozole — ribociclib + letrozole

SUMMARY:
This study was a companion study to CLEE011A2404 which provided the opportunity for the collection of tumor tissue samples to better understand relevant mutations and the mechanisms responsible for resistance to treatment.

DETAILED DESCRIPTION:
This was a multicenter, non-treatment based companion sample collection protocol conducted in the US only. This protocol sought to evaluate the aberrations of common pathways for newly diagnosed HR+/HER2- advanced breast cancer tumors and responses to ribociclib in diverse patient populations. This companion sample collection protocol was available for all US patients enrolled on CLEE011A2404 (CompLEEment-1) and did not alter the planned treatment. Tumor collection required for this study occurred at two time points: at baseline/screening and upon the development of progressive disease as shown in the protocol. Patients eligible for this companion study were required to sign an optional additional consent form at the time of enrolling into the core trial.

After eight patients had consented and samples had been taken, it was determined that the companion study protocol had not been properly initiated or monitored at the sites. This was determined to be a significant GCP violation and the clinical team made the decision to terminate the trial. In addition to the GCP issues, enrollment had been closed to the core study so enrolling additional patients was no longer possible. The limited number of samples would not provide any meaningful analysis. The samples were never analyzed. The study was not terminated due to safety or efficacy concerns. Samples collected were either destroyed or will be retained for up to 15 years based upon the decision of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was to have been obtained prior to any baseline/screening procedures.
* Patients eligible for this companion sample collection protocol sample collection protocol must have met all inclusion in CLEE011A2404.

Exclusion Criteria:

* Patients eligible for this companion sample collection protocol must not have met any of the exclusion criteria in the CLEE011A2404 study, in addition to the following:
* Patients without either fresh or archival tumor tissue accessible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Arizona Oncology Associates PC HAL, Sedona, Arizona
  - Pacific Shores Medical Group SC, Long Beach, California
  - Oncology Speciialists of Charlotte, Charlotte, North Carolina
  - McLeod Center for Cancer Treatment and Research, Florence, South Carolina
  - Carolina Blood and Cancer Care of South Carolina, Rock Hill, South Carolina
  - PeaceHealth St Joseph Medical Center, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients had to have met all eligibility criteria and to have been enrolled into the CLEE011A2404 core study. Patients were offered the opportunity to consent and enroll into this optional companion study.
Groups:
- Ribociclib + Letrozole: ribociclib with letrozole
Period: Overall Study
Arm/Group | Ribociclib + Letrozole
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study terminated by sponsor | 8

BASELINE CHARACTERISTICS:
Arm/Group | Ribociclib + Letrozole
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 6
  Black | 2

OUTCOME MEASURES:

1. Primary Outcome: Identify Mutations of Genes From Tissue Samples Between Baseline and Time to Progression to Determine Modes of Resistance to Ribociclib After Disease Progression
Description: Mutations of genes that were relevant to HR+ and the CDK4/6 pathway such as but not limited to CCND1, CDKN2A, PIK3CA and PTEN to identify the potential mechanisms of progression.
Time Frame: Baseline, time of progression approximately 24 months
Population: No samples were analyzed
Arm/Group | Ribociclib + Letrozole
Number analyzed (Participants) | 0

2. Secondary Outcome: Compare the Differences in Mutations Across Various Races / Ethnicities Based on Baseline Samples
Description: Change in mutations would have been assessed based on baseline samples and compared across diverse races/ethnicities with HR+ HER2- advanced breast cancer - specifically Caucasian, African America, Hispanic, Native American and Pacific Islander.
Time Frame: Baseline, time of progression approximately 24 months
Population: No samples were analyzed
Arm/Group | Ribociclib + Letrozole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First biomarker sample collected up to approximately 21 months biomarker collection procedure SAEs were to have been collected in CORE study (CLEE011A2404)
Description: Only serious adverse events related to biomarker collection procedure were to be collected for this companion study and were to have been reported in CORE study (CLEE011A2404). There were no biomarker collection procedure SAEs reported. All cause mortality and other adverse events were not assessed.
Arm/Group | Ribociclib + Letrozole
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03050398/Prot_SAP_001.pdf